CLINICAL TRIAL: NCT00967668
Title: ASPIRE: Coaching Veterans to Healthy Weights and Wellness
Brief Title: Coaching Veterans to Healthy Weights and Wellness
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IBB 09-034
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-02

CONDITIONS: Obesity
Keywords: Counseling; Veterans; Weight loss; Physical activity; Diet
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ASPIRE-Phone Lifestyle Coaching (Experimental): Phone-based coaching using small change approach to improve physical activity and diet. Initial treatment of 3 months, followed by 21 months of follow-up phone support (phone-only ASPIRE-VA).
  Interventions: Behavioral: Small change approach to improve physical activity and diet
- ASPIRE-Group Lifestyle Coaching (Experimental): On-site weekly group visits using small change approach to improve physical activity and diet. Initial treatment of 3 months, followed by 21 months of follow-up phone support (phone-only ASPIRE-VA).
  Interventions: Behavioral: Small change approach to improve physical activity and diet
- MOVE! Usual Care (Active Comparator): Usual care MOVE!, which consists of weekly on-site group visits that follow MOVE! protocols with unstructured follow-up phone support
  Interventions: Behavioral: MOVE! Usual Care

INTERVENTIONS:
Behavioral: Small change approach to improve physical activity and diet — The "Aspire to Lifelong Health" (ASPIRE) initial treatment program draws on the strengths of traditional lifestyle change and non-dieting weight loss approaches. ASPIRE incorporates CBT elements, problem-solving therapy, and the small change approach from behavioral choice therapy. For the first week in the program, participants use a food diary to track caloric intake and a pedometer to log their daily physical activity (step counts). Baseline information provides a starting point for participants and their Lifestyle Coach to set one small, but potentially permanent, change in daily food choices and physical activity to promote a caloric deficit. Small changes are cumulative over the weeks and the participant makes their own goals within the context of their own lifestyle.
  Arms: ASPIRE-Group Lifestyle Coaching; ASPIRE-Phone Lifestyle Coaching
Behavioral: MOVE! Usual Care — The MOVE! program offers a stepped-care framework of increasingly intensive treatment. A combination of Level 1 (self-management support) and Level 2 (group sessions and/or individual specialty consultation) will be offered to participants as part of usual care.
  Arms: MOVE! Usual Care

SUMMARY:
ASPIRE has completed enrollment of patients at the Ann Arbor and Cleveland Medical Centers in a study that is examining the impact of an innovative approach to weight loss ("Aspiring to Lifelong Health in VA", aka "ASPIRE-VA"). ASPIRE-VA has 3 key features: 1) lifestyle coaches who encourage behavior change through a "small steps" approach; 2) a simplified "Stoplight" diet; and 3) user-friendly "enhanced" pedometers to help participants monitor their physical activity.

DETAILED DESCRIPTION:
Background:

Nearly 78% of Veterans are overweight or obese, imposing a tremendous burden on the Veterans Health Administration (VHA) healthcare system for the treatment of obesity-related chronic disease and disability. While weight management treatment has been implemented in VHA, program data shows low enrollment, participation, and weight loss. Traditional behavioral weight loss trials frequently exclude individuals with multiple chronic health conditions. Additionally, men are less likely than women to participate in these trials. New weight loss approaches may be needed to treat these populations.

Objectives:

To test whether a small-changes intervention (The Aspiring to Lifelong Health Program; aka ASPIRE), delivered in groups or individually via telephone, promotes greater weight loss than standard obesity treatment in a predominantly male, high-risk Veteran population. Data were collected in 2010-13.

Methods:

A three-arm, 12-month randomized pragmatic effectiveness trial was conducted. Participants were recruited from MOVE! referrals and randomly assigned to one of three programs: the 12-month ASPIRE weight loss program delivered 1) individually over the phone (ASPIRE-Phone) or 2) in-person group sessions (ASPIRE-Group); compared to 3) Veteran Health Administration's VHA standard weight loss program, MOVE!. Participants in the ASPIRE arms met with health coaches weekly in months 1-3, bi-weekly in months 4-9, and monthly in months 10-12. Usual care participants met weekly for 12 weeks with limited options for follow-up care. The ASPIRE program had distinct characteristics: 1) the opportunity for most participants to work with one lifestyle coach throughout treatment, 2) an emphasis on behavior change through a "small steps" approach; 3) the prominence of self-monitoring both physical activity and food intake as a weight loss tool; and 4) the addition of a purely phone based option. Assessments that included the collection of weight, waist circumference and lab values, along with questionnaires, were conducted at baseline, 3-months and 12-months. ASPIRE also added a follow-up component to the study, which was offered to patients at their 12-month assessment. For phone and group patients, it consisted of sessions every other month and an assessment at 18 and 24 months. Usual care patients participated in the assessments only.

Phone-based Interviews were conducted shortly after the 3-month assessment with 19 patients in the ASPIRE phone arm and with 16 in the ASPIRE group arm. These interviews were recorded, transcribed and analyzed using NVivo qualitative software to identify themes associated with successful weight loss at 3-month.

Approximately 5% of all phone and group intervention sessions were audio-recorded. An expert rater used a checklist to rate session fidelity. A second rater independently assessed 30% of the recorded sessions to establish inter-rater reliability. The checklist was psychometrically validated. It was hypothesized that greater adherence to core behavioral change processes and patient-centered communication strategies by the interventionists would be associated with higher levels of weight loss.

Using intention-to-treat principles guide all analyses. The primary outcome was weight change and secondary outcomes included changes in anthropometric (e.g., waist circumference), behavioral, fitness, psychosocial, and physiological measures. The primary analytic approach relied on a linear mixed-effects model with baseline, 3- and 12-month outcomes (e.g., weight) as dependent variables, with each subject as a random intercept to adjust for within-patient correlation of the repeated measures, fixed predictors of study arm indicators, 3- and 12-month time indicators, and time-by-study arm interactions.

Status:

All coaching and assessments are complete. A design and rationale paper has been published, a paper highlighting 12-month results is in revision. Papers on fidelity, qualitative findings, the role of mental illness and binge eating on weight loss are in progress. Analyses of 24-month data are underway.

ELIGIBILITY:
Inclusion Criteria:

* Current patient at Ann Arbor or Cleveland medical center.
* Current provider- or self-referral to MOVE! program and eligible to participate in MOVE!
* 18 years of age and older
* Able to communicate in English
* Report being able to walk 10 minutes continuously without sitting down to rest
* Competent to provide written informed consent

Exclusion Criteria:

* Enrolled in another research study involving weight loss, nutrition, or physical activity
* Being treated for weight loss or on weight loss medications (OTC or prescribed)
* Are currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie C Lowery, PhD MHSA, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - VA Medical Center, Cleveland, Cleveland, Ohio

REFERENCES:
- [Result] Lutes LD, Dinatale E, Goodrich DE, Ronis DL, Gillon L, Kirsh S, Richardson CR, Damschroder LJ. A randomized trial of a small changes approach for weight loss in veterans: design, rationale, and baseline characteristics of the ASPIRE-VA trial. Contemp Clin Trials. 2013 Jan;34(1):161-72. doi: 10.1016/j.cct.2012.09.007. Epub 2012 Oct 4. PMID 23041618
- [Result] Damschroder LJ, Lutes LD, Kirsh S, Kim HM, Gillon L, Holleman RG, Goodrich DE, Lowery JC, Richardson CR. Small-changes obesity treatment among veterans: 12-month outcomes. Am J Prev Med. 2014 Nov;47(5):541-53. doi: 10.1016/j.amepre.2014.06.016. Epub 2014 Sep 10. PMID 25217098
- [Derived] Janney CA, Masheb RM, Lutes LD, Holleman RG, Kim HM, Gillon LR, Damschroder LJ, Richardson CR. Mental health and behavioral weight loss: 24-month outcomes in Veterans. J Affect Disord. 2017 Jun;215:197-204. doi: 10.1016/j.jad.2017.03.003. Epub 2017 Mar 11. PMID 28340446
- [Derived] Damschroder LJ, Goodrich DE, Kim HM, Holleman R, Gillon L, Kirsh S, Richardson CR, Lutes LD. Development and validation of the ASPIRE-VA coaching fidelity checklist (ACFC): a tool to help ensure delivery of high-quality weight management interventions. Transl Behav Med. 2016 Sep;6(3):369-85. doi: 10.1007/s13142-015-0336-x. PMID 27528526
- [Derived] Vimalananda V, Damschroder L, Janney CA, Goodrich D, Kim HM, Holleman R, Gillon L, Lutes L. Weight loss among women and men in the ASPIRE-VA behavioral weight loss intervention trial. Obesity (Silver Spring). 2016 Sep;24(9):1884-91. doi: 10.1002/oby.21574. Epub 2016 Aug 4. PMID 27488278
- [Derived] Masheb RM, Lutes LD, Kim HM, Holleman RG, Goodrich DE, Janney CA, Kirsh S, Higgins DM, Richardson CR, Damschroder LJ. Weight loss outcomes in patients with pain. Obesity (Silver Spring). 2015 Sep;23(9):1778-84. doi: 10.1002/oby.21160. Epub 2015 Aug 3. PMID 26237112

RESULTS

PARTICIPANT FLOW:
Groups:
- ASPIRE-Phone Lifestyle Coaching: Phone-based initial treatment of 3 months, followed by 21 months of follow-up phone support (phone-only ASPIRE-VA)
  Small change approach to improving physical activity and diet: The "Aspire to Lifelong Health" (ASPIRE) program is an innovative approach to weight management drawing on the strengths of both traditional lifestyle change and non-dieting weight loss approaches. ASPIRE incorporates CBT elements, problem-solving therapy, and the small change approach from behavioral choice therapy. For the first week participants use a food diary to track food intake and a pedometer to log their physical activity (step counts). Using this baseline information as a starting point, in each subsequent week participants work with a Lifestyle Coach to set small, but potentially permanent, changes in food choices and physical activity that will promote a caloric deficit. These small changes are cumulative and the participant makes their own goals within the context of their own lifestyle.
- ASPIRE-Group Lifestyle Coaching: On-site weekly group visits for 3 months, followed by 21 months of follow-up groups. (on-site ASPIRE-VA)
  Small change approach to improving physical activity and diet: The "Aspire to Lifelong Health" (ASPIRE) program is an innovative approach to weight management drawing on the strengths of both traditional lifestyle change and non-dieting weight loss approaches. ASPIRE incorporates CBT elements, problem-solving therapy, and the small change approach from behavioral choice therapy. For the first week participants use a food diary to track food intake and a pedometer to log their physical activity (step counts). Using this baseline information as a starting point, in each subsequent week participants work with a Lifestyle Coach to set small, but potentially permanent, changes in food choices and physical activity that will promote a caloric deficit. These small changes are cumulative and the participant makes their own goals within the context of their own lifestyle.
Period: Overall Study
Arm/Group | ASPIRE-Phone Lifestyle Coaching | ASPIRE-Group Lifestyle Coaching | MOVE! Usual Care
Started | 162 | 160 | 159
3-mo Assessment | 131 | 127 | 115
Completed Year 1 - 12-mo Assessment | 120 | 122 | 119
18-mo Assessment | 95 | 102 | 92
Completed | 91 | 104 | 90
Not Completed | 71 | 56 | 69
Not completed — Withdrawal by Subject | 13 | 8 | 8
Not completed — Death | 0 | 2 | 4
Not completed — Removed due to behavior | 1 | 1 | 2
Not completed — Refused Year 2 | 11 | 6 | 4
Not completed — Lost to follow-up at 12-mo | 27 | 29 | 26
Not completed — Lost to Follow-up | 15 | 9 | 16
Not completed — Refused 12-mo assessment | 3 | 1 | 9
Not completed — Pregnancy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of participants randomized to each arm
Groups:
- ASPIRE-Phone Lifestyle Coaching: Phone-based initial treatment of 3 months, followed by 21 months of follow-up phone support (phone-only ASPIRE-VA)
  Small change approach to improving physical activity and diet: The "Aspire to Lifelong Health" (ASPIRE) program is an innovative approach to weight management drawing on the strengths of both traditional lifestyle change and non-dieting weight loss approaches. ASPIRE incorporates elements from cognitive behavioral therapy, problem-solving therapy, and behavioral choice therapy. For the first week participants use a food diary to track food intake and a pedometer to log their physical activity (step counts). Using this baseline information as a starting point, in each subsequent week participants work with a Lifestyle Coach to set small, but potentially permanent, changes in food choices and physical activity that will promote a caloric deficit. These small changes are cumulative and the participant makes their own goals within the context of their own lifestyle.
- ASPIRE-Group Lifestyle Coaching: On-site weekly group visits for 3 months, followed by 21 months of follow-up groups. (on-site ASPIRE-VA)
  Small change approach to improving physical activity and diet: The "Aspire to Lifelong Health" (ASPIRE) program is an innovative approach to weight management drawing on the strengths of both traditional lifestyle change and non-dieting weight loss approaches. ASPIRE incorporates elements from cognitive behavioral therapy, problem-solving therapy, and behavioral choice therapy. For the first week participants use a food diary to track food intake and a pedometer to log their physical activity (step counts). Using this baseline information as a starting point, in each subsequent week participants work with a Lifestyle Coach to set small, but potentially permanent, changes in food choices and physical activity that will promote a caloric deficit. These small changes are cumulative and the participant makes their own goals within the context of their own lifestyle.
- Total: Total of all reporting groups
Arm/Group | ASPIRE-Phone Lifestyle Coaching | ASPIRE-Group Lifestyle Coaching | MOVE! Usual Care | Total
Number analyzed (Participants) | 162 | 160 | 159 | 481
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10.0) | 54.9 (9.5) | 54.6 (10.5) | 55.0 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 20 | 72
  Male | 136 | 134 | 139 | 409
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 67 | 65 | 64 | 196
  White | 91 | 94 | 91 | 276
  Other | 4 | 1 | 4 | 9
Education, years [Number; unit: participants]
  Less than 13 | 38 | 34 | 36 | 108
  13-15 | 81 | 81 | 92 | 254
  16 or more | 40 | 42 | 26 | 108
  Missing | 3 | 3 | 5 | 11
Income less than $20k [Number; unit: participants]
  Income less than $20k | 55 | 70 | 71 | 196
  Income $20k or more | 107 | 90 | 88 | 285
Health-related disability [Number; unit: participants]
  Yes | 74 | 87 | 88 | 249
  No | 88 | 73 | 71 | 232
Charlson Index [Mean (Standard Deviation); unit: units on a scale] — * Indicates burden of disease (Ref #1 below).
  * Total score reported. Published score range 0-8 (see Ref #2 below).
  * Lower score indicates lower burden of disease; 1-point increase in score value is approximately 1.45 increase in relative risk of death.
  * Scores computed by assigning "points" based on disease and age (See Ref #2)
  Refs: Quan H, et al. Coding algorithms for defining comorbidities in ICD-9-CM and ICD-10 administrative data. Med Care 2005;43(11):1130-9.
  Charlson M, et al. Validation of a combined comorbidity index. J. Clin. Epidemiol. Nov 1994;47(11):1245-1251.
  units on a scale | 1.0 (1.3) | 1.2 (1.4) | 1.2 (1.6) | 1.1 (1.5)
Depression [Number; unit: participants]
  Yes | 35 | 62 | 59 | 156
  No | 127 | 98 | 100 | 325
Diabetes [Number; unit: participants]
  Yes | 53 | 64 | 60 | 177
  No | 109 | 96 | 99 | 304

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Expected weight change from baseline to 12 months in kilograms based on linear mixed-effects model using all available data
Time Frame: 12 months after enrollment
Measure: Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | ASPIRE-Phone Lifestyle Coaching | ASPIRE-Group Lifestyle Coaching | MOVE! Usual Care
Number analyzed (Participants) | 162 | 160 | 159
Kilograms | -1.4 [-2.4 to -0.5] | -2.8 [-3.8 to -1.9] | -1.4 [-2.3 to -0.4]
Statistical Analysis 1: Comparison: ASPIRE-Phone Lifestyle Coaching vs ASPIRE-Group Lifestyle Coaching vs MOVE! Usual Care; All participants were included in outcomes analyses using intention-to-treat principles. A linear mixed-effects model with baseline, 3- and 12-month outcome values modeled as dependent variables was used.This statistical approach allows the use of data from all participants as long as the dependent variable is available for at least one time point. Each subject was included as a random intercept to adjust for within-person correlations; Test type: Superiority or Other; p < 0.05, Regression, Linear; Linear mixed-effects model with baseline, 3- and 12-month outcome values modeled as dependent variables

2. Secondary Outcome: Change in Weight
Description: Expected weight change from baseline to 24 months in kilograms based on linear mixed-effects model using all available data. Statistical analyses methods are the same as for the 12-month outcome.
Time Frame: 24 months after enrollment
Population: Includes only individuals who formally consented to participate in the second 12 months of the study.
Measure: Mean (95% Confidence Interval); unit: kilograms
Groups:
- Arm 1: Phone-based initial treatment of 3 months, followed by 21 months of follow-up phone support (phone-only ASPIRE-VA)
  Small change approach to improving physical activity and diet: The "Aspire to Lifelong Health" (ASPIRE) program is an innovative approach to weight management drawing on the strengths of both traditional lifestyle change and non-dieting weight loss approaches. ASPIRE incorporates CBT elements, problem-solving therapy, and the small change approach from behavioral choice therapy. For the first week participants use a food diary to track food intake and a pedometer to log their physical activity (step counts). Using this baseline information as a starting point, in each subsequent week participants work with a Lifestyle Coach to set small, but potentially permanent, changes in food choices and physical activity that will promote a caloric deficit. These small changes are cumulative and the participant makes their own goals within the context of their own lifestyle.
- Arm 2: On-site weekly group visits for 3 months, followed by 21 months of follow-up groups. (on-site ASPIRE-VA)
  Small change approach to improving physical activity and diet: The "Aspire to Lifelong Health" (ASPIRE) program is an innovative approach to weight management drawing on the strengths of both traditional lifestyle change and non-dieting weight loss approaches. ASPIRE incorporates CBT elements, problem-solving therapy, and the small change approach from behavioral choice therapy. For the first week participants use a food diary to track food intake and a pedometer to log their physical activity (step counts). Using this baseline information as a starting point, in each subsequent week participants work with a Lifestyle Coach to set small, but potentially permanent, changes in food choices and physical activity that will promote a caloric deficit. These small changes are cumulative and the participant makes their own goals within the context of their own lifestyle.
- Arm 3: Usual care MOVE!, which consists of weekly on-site group visits that follow MOVE! protocols with unstructured follow-up phone support
  MOVE! Usual Care: The MOVE! program offers a stepped-care framework of increasingly intensive treatment. A combination of Level 1 (self-management support) and Level 2 (group sessions and/or individual specialty consultation) will be offered to participants as part of usual care.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 105 | 115 | 112
kilograms | -1.91 [-3.15 to -0.66] | -1.3 [-2.47 to -0.12] | -1.8 [-3.05 to -0.55]

ADVERSE EVENTS:
Time Frame: Adverse events are reported for the full 2-years of participation of each individual.
Description: For every category, events are based on what patients self-reported to a study team member. ASPIRE participants had more opportunities to report events because of interactions with their coach in addition to assessments. MOVE! participants only reported at assessments.
Arm/Group | ASPIRE-Phone Lifestyle Coaching | ASPIRE-Group Lifestyle Coaching | MOVE! Usual Care
Serious Adverse Events (participants affected / at risk) | 0/162 | 0/160 | 0/159
Other Adverse Events (participants affected / at risk) | 45/162 | 33/160 | 15/159
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ASPIRE-Phone Lifestyle Coaching (N=162) | ASPIRE-Group Lifestyle Coaching (N=160) | MOVE! Usual Care (N=159)
sore muscles and joints (Musculoskeletal and connective tissue disorders) | 41 | 24 | 10
stomach problems (Gastrointestinal disorders) | 2 | 0 | 0
multiple systems or other (General disorders) | 3 | 6 | 1
minor injuries while exercising (Injury, poisoning and procedural complications) | 3 | 5 | 0
sinus, breathing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
rashes (Skin and subcutaneous tissue disorders) | 2 | 5 | 1
low pulse, chest pain (Cardiac disorders) | 0 | 1 | 1
blood sugar (Endocrine disorders) | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes